CLINICAL TRIAL: NCT01889953
Title: EUS-Guided Biliary Drainage in Patients With Inoperable Malignant Distal Biliary Obstruction and Failed ERCP: a Prospective Feasibility Multicenter Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Indiana University (Other); University of Colorado, Denver (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); All India Institute of Medical Sciences (Other); Winthrop University Hospital (Other); University of Florida (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Erasmus Medical Center (Other); AdventHealth (Other); Medical University of South Carolina (Other); Institute of advanced endoscopy (Unknown); Aichi Cancer Center (Other)
Responsible Party: Principal Investigator, Mouen Khashab, Assistant Professor of Medicine; Director of Therapeutic Endoscopy, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00077483
Record Dates: First submitted 2012-12-04; First posted 2013-07-01 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-01

CONDITIONS: Malignant Distal Biliary Obstruction
Keywords: EUS-Guided Biliary Drainage; Endoscopic retrograde cholangiopancreatography; Malignant Biliary Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-guided biliary drainage (Other): Patients in this arm will receive EUS-guided biliary drainage.
  Interventions: Other: EUS-guided biliary drainage

INTERVENTIONS:
Other: EUS-guided biliary drainage — Based on the patient's condition, the will receive:
  * Rendezvous technique
  * Direct transluminal access transesophageal technique
  * Direct transluminal access transduodenal technique
  * or direct transluminal access using transgastric approach

SUMMARY:
This research is being done to study the safety and feasibility of recruiting patients eligible for EUS-guided biliary drainage (EGBD). Our goal is to prospectively study safety and effectiveness of this procedure.

DETAILED DESCRIPTION:
Our central hypothesis is that EGBD is equally effective and safe to percutaneous transhepatic biliary drainage (PTBD) but is associated with better quality of life than PTBD in patients with inoperable malignant distal biliary obstruction who have failed prior ERCP. Furthermore, EGBD may be associated with decreased procedure-related costs. Patients who undergo PTBD usually require multiple procedures for stent exchange/upsize. Our initial study will be a prospective multicenter feasibility study that will include patients with inoperable distal biliary obstruction who have failed ERCP. If feasibility is demonstrated, our goal will be to compare EGBD and PTBD in a randomized multicenter international trial with a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (18-80 years of age) with jaundice due to inoperable (by EUS and/or CT criteria or due to health status) malignant distal (more than 2cm distal to hilum) biliary obstruction and who have failed prior ERCP attempt. Failure is considered to be 2 unsuccessful attempts, according to each institution's definition of "failed" procedure (patients may be consented for EGBD prior to repeat ERCP due to higher likelihood of failure). One failure at outside institution and one failure at your institution can be considered as total of two failures.
* Ability to give informed consent

Exclusion Criteria:

* Unable to give informed consent
* Life expectancy < 1month
* Pregnant or breastfeeding women
* Acute gastrointestinal bleeding
* Coagulopathy defined by prothrombin time < 50% of control; PTT > 50 sec, or INR > 1.5), or on chronic anticoagulation
* Inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other contraindication to endoscopy.
* Prior total gastrectomy, Roux-en-Y gastric bypass, esophagectomy and sleeve gastrectomy
* ESLD with portal hypertension, varices, and/or ascites
* Liver metastases burden > 30%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness (Clinical success is defined as drop in bilirubin by 50%) | From date of intervention up to 4 weeks
  Clinical success is defined as drop in bilirubin by 50% at 2 weeks and to below 3 (level

SECONDARY OUTCOMES:
Quality of life (QOL) | From date of intervention up to 12 weeks
  Determine improvement in QOL of patients after PTBD. QOL will be assessed using the EORTC-QLQ-30 instrument (at baseline, 1 week, 4 weeks and 12 weeks after the procedure).
Procedure-related costs | Lifetime (These patients have a life expectancy of less than 2 years)
  Cost will be determined according to Medicare reimbursement of billed CPT codes. The cost of all related follow-up procedures will be included (e.g. cost of PTBD in case of failed EGBD, cost of managing complications, cost of reintervention in case of stent occlusion, etc)
Number of required procedures | From date of intervention up to death (These patients have a life expectancy of less than 2 years)
Technical success | Intra- and post intervention (These patients have a life expectancy of less than 2 years)
  This is defined as success of stent placement in the desired location as determined endoscopically and radiographically.
  In addition, success of each step during EUS will be tracked and recorded (e.g. needle puncture, cholangiography, tract dilation, etc
Stent patency | Lifetime (These patients have a life expectancy of less than 2 years)
  Determine stent patency which is defined as time period between stent placement and need for reintervention for signs and symptoms of recurrent biliary obstruction
Determine safety of EGBD (Complications include the following: Bile leak, Perforation, Peritonitis, Cholecystitis) | Lifetime (These patients have a life expectancy of less than 2 years)
  Complications include the following: Bile leak, Perforation, Peritonitis, Cholecystitis

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins Hospital Department of Gastroenterology
Locations (13):
- United States (7):
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Florida Hospital, Orlando, Florida
  - Indiana University, Bloomington, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Winthrop University Hospital, Mineola, New York
  - Medical University of South Carolina, Charleston, South Carolina
- India (2):
  - All India Institute of Medical Sciences, Delhi
  - Institute of advanced endoscopy, Mumbai
- Ismett/Upmc, Palermo, Italy
- Aichi Cancer Center Hospital, Nagoya, Aichi-ken, Japan
- Netherlands (2):
  - Academic Medical Center of Amsterdam, Amsterdam
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Derived] Khashab MA, Van der Merwe S, Kunda R, El Zein MH, Teoh AY, Marson FP, Fabbri C, Tarantino I, Varadarajulu S, Modayil RJ, Stavropoulos SN, Penas I, Ngamruengphong S, Kumbhari V, Romagnuolo J, Shah R, Kalloo AN, Perez-Miranda M, Artifon EL. Prospective international multicenter study on endoscopic ultrasound-guided biliary drainage for patients with malignant distal biliary obstruction after failed endoscopic retrograde cholangiopancreatography. Endosc Int Open. 2016 Apr;4(4):E487-96. doi: 10.1055/s-0042-102648. Epub 2016 Mar 30. PMID 27092334